CLINICAL TRIAL: NCT01639547
Title: A Randomized, Open-lable, Multicenter, Parallel Group Study to Compare SVR Rate of Pegasys Plus Ribavirin for 48 Weeks vs. 36 Weeks in Patients With Chronic Hepatitis C
Brief Title: Sustained Virological Response (SVR)Rate of Pegasys Plus Ribavirin in Patients With Chronic Hepatitis C
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: early termination due to difficult collection of patients
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, I-Shyan Sheen, Clinical Professor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTC-133
Record Dates: First submitted 2012-06-28; First posted 2012-07-12 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Hepatitis C
Keywords: PEGASYS® PLUS RIBAVIRIN
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEGASYS® plus ROBATROL® for 36 weeks (Experimental)
  Interventions: Drug: Peginterferon alfa-2a plus Ribavirin
- PEGASYS® plus ROBATROL® for 48 weeks (Active Comparator)
  Interventions: Drug: Peginterferon alfa-2a plus Ribavirin

INTERVENTIONS:
Drug: Peginterferon alfa-2a plus Ribavirin — Peginterferon alfa-2a(pre-filled syringes 180 mcg/0.5 ml once a week) plus ribavirin(200 mg/Capsules, 1000~1200 mg daily in split doses (morning/evening)) for 36 or 48 weeks
  Other Names: PEGASYS® plus ROBATROL®

SUMMARY:
The purpose of this study is to evaluate the effect of PEGASYS® (peginterferon alfa-2a 40KD) plus Robatrol® (ribavirin) combination therapy given for 36 weeks versus 48 weeks on the clearance of HCV viremia 24 weeks after treatment end

DETAILED DESCRIPTION:
Pegylated interferon plus ribavirin brings a good therapeutic response and curability. However, the adverse effects and sufferings are lots. Response-guided, personalized treatment is current principle. In patients of CHC, GT1 PR treatment for 24 weeks is established in rapid virologic responders (RVR) who have low viral load before treatment. As to patients with RVR but high viral load (HVL), the treatment duration is 48 weeks that is the same as patients with complete early virologic response (cEVR). Is a shorter duration of treatment feasible for those with a good virokinetic response? The ideal treatment duration for patients of chronic hepatitis C, GT-1, high viral load with RVR has had no enough data yet. Is it really necessary to double the treatment duration (48 weeks) for patients of chronic hepatitis C, GT-1, high viral load with RVR? Is 36-week adequate for them? A multicenter trial of INDIV-2 was presented at EASL 2010. They treated CHC patients of naïve GT1 HVL and RVR for 30 weeks and got similarly good SVR as those treated for 48 weeks (85% vs. 82%).

Therefore, investigators design a randomized controlled study to investigate the SVR rates between treatment for 36 weeks and for 48 weeks in patients of CHC, GT1, HVL and RVR.

ELIGIBILITY:
Inclusion Criteria:

* 20~70 years old
* Patients have never been treated with traditional interferon plus ribavirin or peginterferon plus ribarivin
* Chronic hepatitis C, genotype 1, HCV-RNA > 0.8x106 IU/ml, achieving RVR (undetectable HCV RNA at week 4) in the SoC treatment
* Patient must be able to comply with the assessments during the study
* Compensated liver disease (Child-Pugh Grade A clinical classification for patients with cirrhosis: total score ≦ 6)
* All fertile males and females receiving ribavirin must be using two forms of effective contraception during treatment with study drugs and 6 months post treatment completion

Exclusion Criteria:

* History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures)
* History or other evidence of decompensated liver disease
* Signs or symptoms of hepatocellular carcinoma
* Co-infection with hepatitis A, hepatitis B or human immunodeficiency virus (HIV)
* Not adequately controlled thyroid dysfunction, diabetes mellitus (HbA1c >8.5%) or psychiatric disorders, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at therapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt, hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease
* History of a severe seizure disorder or current anticonvulsant use
* History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study
* Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration) or clinically relevant ophthalmological disorder (e.g. due to diabetes mellitus or hypertension)
* Women with on-going pregnancy or breast feeding
* Male partners of women who are pregnant
* Subjects with any of the following laboratory abnormalities

  * Platelet count < 90,000/mm3
  * Absolute neutrophil count < 1,500 /mm3
  * Hemoglobin < 12 g/dL (F), 13 g/dL (M)
  * Creatinine > ULN
  * ALT and/or AST > 10X ULN
  * Total serum bilirubin > 1.5 x ULN
* Inability or unwillingness to provide written informed consent or abide by the requirements of the study

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | At 24 weeks after end of treatment
  Sustained virological response (SVR) defined as percentage of patients with HCV RNA < 15 IU/ML as measured by the Roche COBAS AmpliPrep / COBAS TaqMan® HCV Test at 24 weeks post completion of the 36 or 48 week treatment periods.

SECONDARY OUTCOMES:
Virological Response Rate at week 2 | At treatment week 2
  Virological Response Rate at week 2 defined as the percentage of patients with HCV RNA < 15 IU/ML as measured by the Roche COBAS AmpliPrep / COBAS TaqMan® HCV at 2 weeks post treatment.
Virological response at end of treatment | At end of treatment
  Virological response at end of treatment defined as the percentage of patients with HCV RNA < 15 IU/ML as measured by the Roche COBAS AmpliPrep / COBAS TaqMan® HCV Test after the last dose of study medication(± 28 days).
Correlation of virological response and SVR rate | At 24 weeks after end of treatment
  Correlation of virological response (HCV RNA < 15 IU/ML) at week 2 and SVR rate in each group.

CONTACTS AND LOCATIONS:
Overall Officials: I-Shyan Sheen, M.D., Principal Investigator — Linkou Medical Center, Chang Gung Memorial Hospital
Locations (7):
- Taiwan (7):
  - Show Chwan Memorial Hospital, Changhua
  - Changhua Christian Hospital, Changhua County
  - Keelung Chang Gung Memorial Hospital, Keelung
  - China Medical University Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - Taipei Medical University - Shuang Ho Hospital, Taipei County
  - Linkou Medical Center, Chang Gung Memorial Hospital, Taoyuan